CLINICAL TRIAL: NCT03299426
Title: A Phase III Randomized, Double-Blind, Controlled Trial of the Clinical Efficacy of Typhoid Conjugate Vaccine (Vi-TCV) Among Children Age 9 Months Through 12 Years in Blantyre, Malawi
Brief Title: Clinical Efficacy of Typhoid Conjugate Vaccine (Vi-TCV) Among Children Age 9 Months Through 12 Years in Blantyre, Malawi
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); University College, London (Other); University of Malawi (Other)
Responsible Party: Principal Investigator, Matthew Laurens, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HP-00076625
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Typhoid
Keywords: Typhoid; Typhoid in Malawi; Typhoid Vaccine
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vi-Typhoid Conjugate Vaccine (Vi-TCV) (Experimental): Children will receive a single 0.5-ml dose of Vi-TCV administered by the intramuscular route.
  Interventions: Biological: Vi-Typhoid Conjugate Vaccine (Vi-TCV)
- Meningococcal A Conjugate Vaccine (MCV-A) (Active Comparator): Children will receive a single dose of MCV-A administered by the intramuscular route. Children 9-11 months will receive a 5µg/0.5ml dose. Children 12 months and older will receive a 10µg/0.5 ml dose.
  Interventions: Biological: Meningococcal A Conjugate Vaccine (MCV-A)

INTERVENTIONS:
Biological: Vi-Typhoid Conjugate Vaccine (Vi-TCV) — Single 0.5-ml intramuscular injection
  Arms: Vi-Typhoid Conjugate Vaccine (Vi-TCV)
Biological: Meningococcal A Conjugate Vaccine (MCV-A) — Single intramuscular injection. Children 9-11 months will receive a 5µg/0.5ml dose. Children 12 months and older will receive a 10µg/0.5 ml dose.
  Arms: Meningococcal A Conjugate Vaccine (MCV-A)

SUMMARY:
This study will evaluate the efficacy of a Typhoid conjugate vaccine (Vi-TCV) in Malawi, Africa among children age 9 months through 12 years. Participants will be randomized in a 1:1 ration to receive the study vaccine or the control vaccine (meningococcal group A conjugate vaccine - MCV-A).

DETAILED DESCRIPTION:
This study is a double-blind, individually randomized, controlled, clinical efficacy trial with two vaccine groups: Vi-TCV (Typhoid conjugate) and MCV-A (meningococcal group A conjugate). This study will take place in Blantyre, Malawi, Africa. Participants (up to 30,000) will be randomized in a 1:1 ratio. Children 9 months through 12 years of age in the Blantyre area who meet the inclusion criteria will be eligible for enrollment.

Participants will be unaware of which study vaccine, Vi-TCV or MCV-A, is received. A subset of 600 children will have study visits on days 3, 7, 28 and 180 post-vaccination to assess select solicited events, unsolicited events, and all serious adverse events. Serious Adverse Events (SAEs) in all participants will be monitored through the end of the trial.

For the evaluation of efficacy, passive surveillance will be conducted for up to 36 months to identify cases among vaccinated subjects. Children who meet the protocol-defined specimen collection criteria will have a blood culture collected. Additional information will be collected from any child who has a blood culture obtained. This will include information about the signs and symptoms of the illness and treatment given. Likewise, any child with blood culture-confirmed typhoid fever will have follow-up until the illness resolves. Additional information on the illness, treatment and complications will be recorded. Vaccine efficacy will be evaluated when the pre-specified number of cases is reached after a minimum of two years of follow-up on each participant.

A subset of 600 children (200 in each of three age groups: 9-11 months, 1-5 years, and 6-12 years) will be included in an additional Vaccine Immunogenicity and Reactogenicity Sub-study. More stringent exclusion criteria will apply for this subset. The purpose of this detailed evaluation is to assess the reactogenicity of the vaccine and the immune responses to Vi-TCV. Serum specimens will be collected on day 0 (before vaccination) and on post-vaccination days 28 and 730 from all children included in the sub-study. For the children in the 9-11 month group, Vi-TCV or MCV-A will be administered with measles-containing vaccine, as per Malawi Expanded Programme on Immunization (EPI) schedule. These 9-11-month-old children will have antibody to measles assessed on days 0 and 28. All children in the sub-study will have visits at days 4 and 7 following vaccination for solicitation of local and systemic adverse events. Serious and non-serious adverse events will be assessed at days 28 and 180.

An additional subset of -up to 225 HIV-exposed-but-uninfected and up to 100 HIV-unexposed children ages 9-11 months will be included in an additional HIV-exposed Vaccine Immunogenicity and Reactogenicity Substudy. The purpose of this detailed evaluation is to assess the reactogenicity of the vaccine and the immune responses to one or two doses of Vi-TCV in HIV-exposed children. Up to 225 HIV-exposed children in this substudy will be randomized 1:1:1 to receive either TCV at 9-11 months and TCV at 15 months (Group 1), TCV at 9-11 months only (Group 2), or TCV at 15 months only (Group 3). A separate group of about 100 HIV-unexposed children will serve as controls and receive TCV at 9-11 months and TCV at 15 months (Group 4). Serum specimens will be collected on day 0 (before vaccination) and on 28 days after each vaccination from all children included in the sub-study. For this substudy, Vi-TCV will be administered with measles-rubella-containing vaccine #1 at 9-11 months and/or #2 at 15 months, as per Malawi EPI schedule. These 9-11-month-old children will have antibody to typhoid, measles, and rubella assessed on day 0 and 28 days after each vaccination. All children in the sub-study will be assessed at 7 days after each vaccination for solicitation of local and systemic adverse events. Serious and non-serious adverse events will be assessed up to the last study visit for HIV-exposed substudy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female child between the ages of 9 months and 12 years/364 days at the time of study vaccination.
* A child whose parent or guardian resides primarily within the Ndirande or Zingwangwa study areas at the time of study vaccinations and who intends to be present in the area for the duration of the trial.
* A child whose parent or guardian has voluntarily given informed consent.

Exclusion Criteria:

* History of documented hypersensitivity to any component of the vaccine
* Prior receipt of any typhoid vaccine in the past 3 years
* History of severe allergic reaction with generalized urticarial, angioedema, or anaphylaxis
* Any condition determined by the investigator to be likely to interfere with evaluation of the vaccine or to be a significant potential health risk to the child or make it unlikely that the child would complete the study.

Temporary Exclusion Criteria:

The following will be considered temporary contraindications to enrollment and vaccination. If these apply, the participant will be temporarily excluded for vaccination until 48 hours has passed. A re-assessment will be needed to ensure these temporary exclusion criteria no longer exist.

* Reported fever within 24 hours prior to vaccination
* Use of anti-pyretics within 4 hours prior to vaccination

An additional temporary exclusion criteria will be:

- Receipt of measles vaccine in the one month prior to enrollment, as determined by parental history or vaccination card.

Additional Exclusion Criteria for Safety and Immunogenicity Substudy:

In addition to the exclusion criteria of the efficacy study, participants enrolled in the immunogenicity and reactogenicity substudy may not have, or have had, any:

* Known history of diabetes, tuberculosis, cancer, chronic kidney, heart, or liver disease, progressive neurological disorders, poorly controlled seizures, or terminal illness
* Severe malnutrition as determined by MUAC< 12.5 cm for children younger than 5 years;
* Receipt of any other investigational intervention in the last 6 months or anticipated during the course of the study.
* Receipt of blood products in the last 6 months.
* Known HIV-infection or exposure or other immunosuppressive conditions.
* Receipt of systemic immunosuppressant or systemic corticosteroids.
* Receipt of any measles-containing vaccine for children younger than 1 year of age

Ages: 9 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30000 (Estimated)
Dates: Start 2018-02-21 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Vi-TCV | Up to 36 months
  The primary outcome of interest is the incidence of blood culture-positive typhoid fever among Vi-TCV and MCV-A vaccine recipients in the study population during the entire post-vaccination surveillance period. Vaccine efficacy will be calculated as one minus the relative rate of symptomatic typhoid fever in the Vi-TCV group compared to that in the MCV-A group.

SECONDARY OUTCOMES:
Safety of Vi-TCV | 6 months
  The safety profile of Vi-TCV will be measured by comparing the proportions of participants experiencing solicited and unsolicited local and systemic reactions between children receiving Vi-TCV as compared to children receiving MCV-A according to the following three categories:
  1. The proportion of participants who develop adverse events detected in the first 30 minutes after vaccination and for 7 days after vaccination.
  2. The proportion of participants who experience serious adverse events within 6 months of vaccination in a subset of participants.
  3. The proportion of participants who experience other non-serious adverse events up to 28 days following vaccination, in a subset of participants.
Immunogenicity of Vi-TCV | 28 days
  The immunogenicity of Vi-TCV in a subset of 600 participants measured by ELISA for anti-Vi percent seroconversion and GMTs before and at day 28 after vaccination.
Number of typhoid fever cases prevented Vi-TCV | Up to 36 months
  The number of blood culture-confirmed cases of typhoid fever prevented by Vi-TCV during the study period measured by comparing the incidence of blood culture-confirmed typhoid fever in participants receiving Vi-TCV compared to those receiving MCV-A.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Laurens, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Malawi Liverpool Wellcome Trust Clinical Research Programme, Queen Elizabeth Central Hospital College of Medicine, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel PD, Liang Y, Meiring JE, Chasweka N, Patel P, Misiri T, Mwakiseghile F, Wachepa R, Banda HC, Shumba F, Kawalazira G, Dube Q, Nampota-Nkomba N, Nyirenda OM, Girmay T, Datta S, Jamka LP, Tracy JK, Laurens MB, Heyderman RS, Neuzil KM, Gordon MA; TyVAC team. Efficacy of typhoid conjugate vaccine: final analysis of a 4-year, phase 3, randomised controlled trial in Malawian children. Lancet. 2024 Feb 3;403(10425):459-468. doi: 10.1016/S0140-6736(23)02031-7. Epub 2024 Jan 25. PMID 38281499
- [Derived] Nampota-Nkomba N, Nyirenda OM, Khonde L, Mapemba V, Mbewe M, Ndaferankhande JM, Msuku H, Masesa C, Misiri T, Mwakiseghile F, Patel PD, Patel P, Johnson-Mayo I, Pasetti MF, Heyderman RS, Tracy JK, Datta S, Liang Y, Neuzil KM, Gordon MA, Laurens MB; Typhoid Vaccine Acceleration Consortium team. Safety and immunogenicity of a typhoid conjugate vaccine among children aged 9 months to 12 years in Malawi: a nested substudy of a double-blind, randomised controlled trial. Lancet Glob Health. 2022 Sep;10(9):e1326-e1335. doi: 10.1016/S2214-109X(22)00275-3. PMID 35961356
- [Derived] Patel PD, Patel P, Liang Y, Meiring JE, Misiri T, Mwakiseghile F, Tracy JK, Masesa C, Msuku H, Banda D, Mbewe M, Henrion M, Adetunji F, Simiyu K, Rotrosen E, Birkhold M, Nampota N, Nyirenda OM, Kotloff K, Gmeiner M, Dube Q, Kawalazira G, Laurens MB, Heyderman RS, Gordon MA, Neuzil KM; TyVAC Malawi Team. Safety and Efficacy of a Typhoid Conjugate Vaccine in Malawian Children. N Engl J Med. 2021 Sep 16;385(12):1104-1115. doi: 10.1056/NEJMoa2035916. PMID 34525285
- [Derived] Meiring JE, Laurens MB, Patel P, Patel P, Misiri T, Simiyu K, Mwakiseghile F, Tracy JK, Masesa C, Liang Y, Henrion M, Rotrosen E, Gmeiner M, Heyderman R, Kotloff K, Gordon MA, Neuzil KM. Typhoid Vaccine Acceleration Consortium Malawi: A Phase III, Randomized, Double-blind, Controlled Trial of the Clinical Efficacy of Typhoid Conjugate Vaccine Among Children in Blantyre, Malawi. Clin Infect Dis. 2019 Mar 7;68(Suppl 2):S50-S58. doi: 10.1093/cid/ciy1103. PMID 30845320